CLINICAL TRIAL: NCT03695887
Title: A Pilot Randomized Controlled Crossover Trial of the Effectiveness of Disposable Nitrous Oxide Canisters in Providing Improved Pain Control During Burn Dressing Changes.
Brief Title: A Pilot Trial of Disposable Nitrous Oxide Canisters in Providing Pain Control During Burn Dressing Changes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Sarvesh Logsetty, Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: nitrousoxide
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Burns; Pain, Acute
Keywords: burns, pain, dressing change, nitrous oxide
MeSH Terms: conditions — Burns; Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized to receive either active study article or inactive comparator then crossed over to other treatment arm on next dressing change.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrous Oxide Inhalant Product (Experimental): Nitrous oxide
  Interventions: Drug: Nitrous Oxide Inhalant Product
- Placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrous Oxide Inhalant Product — Nitrous Oxide Inhalant Product
  Arms: Nitrous Oxide Inhalant Product
Drug: Placebo — Inactive comparator
  Arms: Placebo

SUMMARY:
Improvements in burn care have resulted in increased survival. Despite these improved outcomes one of the leading challenges of burn care remains providing adequate analgesia during routine wound care and dressing changes. The traditional use of narcotics is challenging as the therapeutic window between analgesia and suppression of breathing becomes narrow with the intense pain and high doses of narcotics needed for dressing changes.

DETAILED DESCRIPTION:
The normal challenges of using narcotics are increased in burn patients, who have significantly altered metabolism. Unfortunately, the use of regular general anesthesia or conscious sedation is not a viable option due to the resources required, and as the hypermetabolism of burn injury would result in compromised wound healing with repeated periods of without eating related halting of nutritional intake. This has led to the use of a number of adjuncts ranging from nonmedical (virtual reality, mindfulness, hypnosis etc.) to medication (ketamine, anxiolytics etc.). Historically Nitrous oxide has been used in similar settings where severe procedural pain is of relatively shorter duration, such as tooth extraction, labor or minor surgical procedures. Nitrous oxide is a rapidly acting analgesic that takes effect seconds after inhalation, and lasts minutes. While a randomized trial of Nitrous oxide in burn care has been proposed, the only published information currently available is in a Chinese medical journal.

To address this a gap in knowledge, a pilot Randomized Controlled trial is proposed to evaluate if Nitrous Oxide in the form of limited dose inhaler canisters can be used to improve pain control during burn dressing changes compared to placebo canisters.

ELIGIBILITY:
Inclusion criteria

* adult burn patients admitted to the Health Sciences Centre
* total body surface area burned of 5-20%

Exclusion criteria

* admitted to intensive care unit
* unable to participate in the measurement outcomes (sedated, cognitively impaired, unable to understand English or visually impaired)
* medical condition that precludes using nitrous oxide (respiratory disease and significant cardiovascular disease 5).
* pregnant
* physically unable to hold the canister
* <90% SaO2 on room air
* face burn
* pre-injury narcotics (relative exclusion)
* use of IV ketamine
* pre-existing lung injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Burn Specific Pain Anxiety Scale | 1 hour before dressing change
  The experience of the dressing change for the patient will also be assessed using the Burn specific pain and anxiety scale which consists of:
  1. Worry about wound-healing
  2. Fear of procedural pain
  3. Fear of losing control because of pain
  4. Fear of pain during dressing change
  5. Pain severity
  6. Keyed up because of enduring pain
  7. Concern about wound healing
  8. Preoccupied with pain
  9. Tension during dressing change
  Responses for each item are on a visual analogue scale ranging from "least" to "most". The response is normalized to a value between 0 and 1, representing the location selected on the line, divided by the total length of the line. The responses will be used to examine a possible relationship procedural and non procedural pain between the nurse and the patient.
Burn Specific Pain Anxiety Scale | during dressing change
  The experience of the dressing change for the patient will also be assessed using the Burn specific pain and anxiety scale which consists of:
  1. Worry about wound-healing
  2. Fear of procedural pain
  3. Fear of losing control because of pain
  4. Fear of pain during dressing change
  5. Pain severity
  6. Keyed up because of enduring pain
  7. Concern about wound healing
  8. Preoccupied with pain
  9. Tension during dressing change
  Responses for each item are on a visual analogue scale ranging from "least" to "most". The response is normalized to a value between 0 and 1, representing the location selected on the line, divided by the total length of the line. The responses will be used to examine a possible relationship procedural and non procedural pain between the nurse and the patient.
Burn Specific Pain Anxiety Scale | 1 hour after dressing change
  The experience of the dressing change for the patient will also be assessed using the Burn specific pain and anxiety scale which consists of:
  1. Worry about wound-healing
  2. Fear of procedural pain
  3. Fear of losing control because of pain
  4. Fear of pain during dressing change
  5. Pain severity
  6. Keyed up because of enduring pain
  7. Concern about wound healing
  8. Preoccupied with pain
  9. Tension during dressing change
  Responses for each item are on a visual analogue scale ranging from "least" to "most". The response is normalized to a value between 0 and 1, representing the location selected on the line, divided by the total length of the line. The responses will be used to examine a possible relationship procedural and non procedural pain between the nurse and the patient.
Visual Analogue Scale for pain | 1 hour before dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("No pain") and 100 ("worst possible pain").
Visual Analogue Scale for pain | during dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("No pain") and 100 ("worst possible pain").
Visual Analogue Scale for pain | 1 hour after dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("No pain") and 100 ("worst possible pain").
Visual Analogue Scale for anxiety | 1 hour before dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("no anxiety") and 100 ("worst possible anxiety").
Visual Analogue Scale for anxiety | during dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("no anxiety") and 100 ("worst possible anxiety").
Visual Analogue Scale for anxiety | 1 hour after dressing change
  The items are scored on a 100 mm visual analog line with two reference points given values of 0 ("no anxiety") and 100 ("worst possible anxiety").

SECONDARY OUTCOMES:
Anxiolytic given | 1 hour before dressing change
  The amount of anxiolytic given one hour prior to the dressing change.
Anxiolytic given | during dressing change
  The amount of anxiolytic given during the dressing change.
Anxiolytic given | 1 hour after dressing change
  The amount of anxiolytic given one hour after the dressing change.

OTHER OUTCOMES:
Systolic blood pressure | 5 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, systolic blood pressure will be measured.
Systolic blood pressure | 10 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, systolic blood pressure will be measured.
Systolic blood pressure | 15 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, systolic blood pressure will be measured.
Systolic blood pressure | 20 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, systolic blood pressure will be measured.
Diastolic blood pressure | 5 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, Diastolic blood pressure will be measured.
Diastolic blood pressure | 10 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, Diastolic blood pressure will be measured.
Diastolic blood pressure | 15 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, Diastolic blood pressure will be measured.
Diastolic blood pressure | 20 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, Diastolic blood pressure will be measured.
Mean arterial pressure | 5 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, mean arterial pressure (mmHg) will be measured.
Mean arterial pressure | 10 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, mean arterial pressure (mmHg) will be measured.
Mean arterial pressure | 15 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, mean arterial pressure (mmHg) will be measured.
Mean arterial pressure | 20 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, mean arterial pressure (mmHg) will be measured.
Heart rate | 5 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, heart rate will be measured.
Heart rate | 10 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, heart rate will be measured.
Heart rate | 15 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, heart rate will be measured.
Heart rate | 20 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, heart rate will be measured.
Oxygen saturation | 5 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, oxygen saturation will be measured.
Oxygen saturation | 10 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, oxygen saturation will be measured.
Oxygen saturation | 15 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, oxygen saturation will be measured.
Oxygen saturation | 20 minute mark during burn dressing change
  After administration of inhaled nitrous oxide, oxygen saturation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sarvesh Logsetty, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregoretti C, Decaroli D, Piacevoli Q, Mistretta A, Barzaghi N, Luxardo N, Tosetti I, Tedeschi L, Burbi L, Navalesi P, Azzeri F. Analgo-sedation of patients with burns outside the operating room. Drugs. 2008;68(17):2427-43. doi: 10.2165/0003495-200868170-00003. PMID 19016572
- [Background] Yuxiang L, Lu T, Jianqiang Y, Xiuying D, Wanfang Z, Wannian Z, Xiaoyan H, Shichu X, Wen N, Xiuqiang M, Yinsheng W, Ming Y, Guoxia M, Guangyi W, Wenjun H, Zhaofan X, Hongtai T, Jijun Z. Analgesia effect of a fixed nitrous oxide/oxygen mixture on burn dressing pain: study protocol for a randomized controlled trial. Trials. 2012 May 24;13:67. doi: 10.1186/1745-6215-13-67. PMID 22624697
- [Background] Li YX, Tang HT, Zhou WF, Hu XY, Xiao SC, Niu XH, Li YC, Wu YS, Yao M, Wang HX, Xia ZF, Zhao JJ. [Analgesic and sedative effects of inhaling a mixture of nitrous oxide and oxygen on burn patient during and after dressing change]. Zhonghua Shao Shang Za Zhi. 2013 Dec;29(6):537-40. Chinese. PMID 24495641
- [Background] Taal LA, Faber AW, van Loey NE, Reynders CL, Hofland HW. The abbreviated burn specific pain anxiety scale: a multicenter study. Burns. 1999 Sep;25(6):493-7. doi: 10.1016/s0305-4179(99)00034-0. PMID 10498356
- [Background] Becker DE, Rosenberg M. Nitrous oxide and the inhalation anesthetics. Anesth Prog. 2008 Winter;55(4):124-30; quiz 131-2. doi: 10.2344/0003-3006-55.4.124. PMID 19108597